CLINICAL TRIAL: NCT02617264
Title: Spot tm Tattooing of Biopsied Axillary Lymph Nodes With Ultrasound Guided in Breast Cancer Patients Prior to Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Tanir M Allweis, MD, Head of Department of Breast Health Center, Kaplan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KaplanMC
Record Dates: First submitted 2015-10-26; First posted 2015-11-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axillary lymph node FNA Biopsy (Experimental): A carbon compound ink (SPOT) is injected to the axillary lymph node suspected to be infected with cancer
  Interventions: Procedure: SPOT

INTERVENTIONS:
Procedure: SPOT — Injecting the ink (SPOT) to the axillary lymph node prior the surgery. During the surgery the lymph nodes will be tasted to diagnose the marked node.

SUMMARY:
To assess feasibility and clinical utility of marking biopsied axillary lymph nodes with Spot at time of biopsy.

DETAILED DESCRIPTION:
As part of the diagnostic tests for breast cancer sometimes necessary to perform a FNA or Core biopsy to a suspicious axillary lymph node.

Presently there is no possibility to identify the examined gland at the surgery. If the gland was infected it's most important to remove it.

The only technique that exists today is marking with a metal clip and the use of this technique is not profit, partly because of technical difficulties.

In this trial the investigator will use a special ink which will be injected to the axillary lymph node during the biopsy and latter on the surgery the investigator will try to assess the ability to identify the marked gland.

ELIGIBILITY:
Inclusion Criteria:

* Women with findings suspicious of breast cancer (or known breast cancer) who undergo axillary lymph node biopsy

Exclusion Criteria:

* Inability to sign Informed Consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Intra operative identification the Spot TM marked node at the time of surgery | Within 1 year of enrollment

SECONDARY OUTCOMES:
Correlation between Spot TM marked lymph node and sentinel lymph node | Within 1 year of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Tanir Allweis, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Kaplan Medical Center, Rehovot, Israel